CLINICAL TRIAL: NCT06742073
Title: Histiocytosis and Inflammatory Manifestations in Patients with H Syndrome- a Multinational Collaboration
Brief Title: Histiocytosis and Inflammatory Manifestations in Patients with H Syndrome
Status: Recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-0230-24
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: H Syndrome
Keywords: SLC29A3
MeSH Terms: conditions — Histiocytosis with joint contractures and sensorineural deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
H syndrome is a rare genetic disorder predisposing to histiocytosis. Our knowledge of the clinical spectrum of these patients is based on case reports and small patient series. Patients with H syndrome have been treated with a range of immunomodulatory and chemotherapeutic agents, with limited success. We aim to comprehensively assess the clinical manifestations and patterns of treatment response in a multinational cohort of patients with H syndrome.

DETAILED DESCRIPTION:
H syndrome is a rare inflammatory genetic disorder predisposing to histiocytosis, caused by germline biallelic loss-of-function mutations in SLC29A3, encoding the protein equilibrative nucleoside transporter 3 (ENT3). ENT3 transports nucleosides from lysosomes to the cytoplasm following lysosomal degradation of nucleic acids. Results from our previous study (under review) suggest a model in which impaired nucleoside trafficking aberrantly activates nucleoside-sensing Toll-like receptors, leading to persistent activation of ERK, driving histiocytosis. This constitutes a novel signaling pathway leading to activation of ERK and histiocytosis, in the absence of somatic mutations in MAPK cascade genes. Our knowledge of the heterogenous clinical spectrum of these patients is based on case reports and small patient series. Patients with H syndrome have been treated with a range of immunomodulatory and chemotherapeutic agents, with limited success. Improvement following therapy with tocilizumab, an IL6-receptor antibody, has recently been reported in isolated case reports. There is a lack of data on MEK inhibitor therapy in these patients. We aim to comprehensively assess the clinical manifestations and patterns of treatment response in a multinational cohort of patients with H syndrome.

ELIGIBILITY:
Inclusion Criteria: Any patient with a genetically confirmed diagnosis of H syndrome -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a genetically confirmed diagnosis of H syndrome (two pathogenic or likely pathogenic germline SLC29A3 variants)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Response to therapy | 6 months
  complete response/partial response/stable disease/progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Elitzur, MD, Study Director — Schneider Children'ds Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No